CLINICAL TRIAL: NCT06522880
Title: Cytomegalovirus (CMV) Transmission and Immune Tracking (TransmIT) Study: An Observational Study to Evaluate CMV Transmission and Immune Correlates of Viral Shedding Among Young Children in Early Education and Care Settings
Brief Title: Cytomegalovirus (CMV) Transmission and Immune Tracking (TransmIT) Study
Status: Recruiting | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Principal Investigator, Laura Gibson, Professor, University of Massachusetts, Worcester
Other Study IDs: IRB 00000521
Record Dates: First submitted 2024-07-09; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Cytomegalovirus Infections
Keywords: cytomegalovirus; CMV; congenital cytomegalovirus; cCMV
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Children up to and including 36 months in large group childcare centers in the study network
  Interventions: Diagnostic Test: CMV PCR on saliva
- Staff: All staff members in large group childcare centers attended by children participants
  Interventions: Diagnostic Test: CMV PCR on saliva

INTERVENTIONS:
Diagnostic Test: CMV PCR on saliva — Observational study to measure prevalence of CMV shedding by saliva PCR

SUMMARY:
The goal of STAGE I of the CMV TransmIT Study is to determine the prevalence of CMV shedding in children up to and including 36 months of age in large group childcare centers and in staff who regularly work at the center. Participants will complete a health survey and provide one saliva sample for CMV PCR testing. In addition, infrastructure for the study will be developed (e.g. community engagement to build the network of centers, data pipelines, digital platform, sampling workflows) and participant sample collection at home will be piloted. These activities will inform the design of STAGE II.

ELIGIBILITY:
Inclusion Criteria

Children

1. All children up to and including 36 months at time of signed consent regardless of duration of attendance at the center. Children living in the same household can each be enrolled.
2. Parent(s) has provided written informed consent for the child to be screened for CMV by saliva PCR collected at the center or at home

Center Staff

1. Individuals who regularly (average >/= 5 weeks per year) work inside the center in any role, including employed, contracted, volunteer, and full or part time.
2. Staff member has provided written informed consent to be screened for CMV by saliva PCR collected at the center or at home

Exclusion Criteria

Children

1. >/= 37 months of age
2. State Department of Children and Families (DCF) custody

Center Staff

1. Do not regularly (average < 5 days per year) work inside the center
2. Work associated with but not regularly inside the center (e.g. bus drivers or food delivery staff)

Ages: 1 Day to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study participants will be recruited from all children and all staff at each center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of CMV shedding | Stage I up to 2 years
  Prevalence of CMV shedding in children and childcare center staff. Shedding measured by CMV PCR on saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gibson, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States